CLINICAL TRIAL: NCT06943183
Title: Correlation of Gross Motor Movement, and Balance With Screen Time in Healthy Children
Status: Not yet recruiting | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/RCR/AHS/24/0730
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Healthy Children
Keywords: Gross motor movement; balance; screen time; school-aged children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy children: The healthy children group will include school-aged children between 7 to 10 years with no known neurological, musculoskeletal, or developmental disorders. All participants will have normal cognitive function (MMSE ≥ 26) and PBS scores above 20, indicating mild or no motor difficulties.

SUMMARY:
Gross motor function involves large muscle control for activities like walking, running, and sports, and is essential for balance and coordination. Excessive screen time may hinder gross motor development by reducing physical activity, affecting strength and coordination. Structured activities like free play and exercise are key to minimizing these effects. A cross-sectional study will be conducted over 10 months in public and private schools in Lahore. Children aged 7-10 will be included. Screen time will be assessed through demographic data, and gross motor skills evaluated using the TGMD-2. Exclusion criteria: PBS < 20, TGMD-2 < 30, recent orthopedic surgery, and MMSE < 26. Data will be analyzed in SPSS v25 using descriptive statistics and correlation. This study explores the impact of screen time on children's physical development, particularly gross motor skills and balance

DETAILED DESCRIPTION:
This study aims to examine the impact of screen time on gross motor development in school-aged children. Gross motor function, which involves large muscle control for activities such as walking, running, and sports, plays a vital role in developing balance, coordination, and overall physical health. With increased screen use among children, physical activity levels may decrease, potentially affecting their motor development.

A cross-sectional study will be conducted over 10 months in public and private schools across Lahore. The target population includes children aged 7 to 10 years. Screen time exposure will be recorded through demographic questionnaires, and gross motor skills will be assessed using the Test of Gross Motor Development-Second Edition (TGMD-2). Children will be excluded if they have a Pediatric Balance Scale (PBS) score below 20, a TGMD-2 score below 30, recent orthopedic surgery, or a Mini-Mental State Examination (MMSE) score below 26. Data will be analyzed using SPSS version 25 with descriptive statistics and correlation tests. This study seeks to identify how screen time may influence key aspects of children's physical development, particularly focusing on gross motor skills and balance

ELIGIBILITY:
Inclusion Criteria:

* Children between ages 7 to 10 years
* Children with screen time exposure of more than 2 hours per day on a weekday (30,
* Screen time exposure through television, smartphones, tablets, laptops or computers.
* Children with exposure of screen time more than 3 hours on a weekend

Exclusion Criteria:

* Children with Pediatric balance score: below 45.
* Children with TGMD-2 Score: below 30 (less than 10" percentile).
* Children who have had orthopedic surgery within the previous 6 months.
* Cognition Score below 26 on MMSE (Mini-Mental State Examination).

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will consist of children aged 7 to 10 years enrolled in public and private schools in Lahore. Participants must be able to follow basic instructions and engage in physical tasks required for assessment. Children with a Pediatric Balance Scale (PBS) score below 20, TGMD-2 score below 30, a history of orthopedic surgery within the past 6 months, or a Mini-Mental State Examination (MMSE) score below 26 will be excluded. The sample will represent typically developing school-aged children with varying levels of screen time exposure
Sampling Method: Non-Probability Sample
Enrollment: 429 (Estimated)
Dates: Start 2025-04-16 (Estimated); Primary Completion 2025-07-16 (Estimated); Study Completion 2025-07-16 (Estimated)

PRIMARY OUTCOMES:
PBS (Pediatric Berg Balance Scale) | baseline
  The Pediatric Balance Scale (PBS) is a modified version of Berg's Balance Scale, designed for school-aged children with mild to moderate motor difficulties. In a study by Bal et al., 20 children (ages 5-15) with balance disorders were tested twice by the same examiner. Additionally, 10 pediatric physical therapists, unaware of the study hypotheses, rated 10 randomly chosen sessions. The PBS showed excellent reliability, with high test-retest (ICC = 0.998) and interrater (ICC = 0.997) consistency, confirming its effectiveness as a reliable balance assessment tool for this population
Screen Time Questionnaire | baseline
  The Pediatric Balance Scale (PBS), a modified Berg's Balance Scale, is for school-aged children with mild to moderate motor difficulties. In a study by Bal et al., 20 children (ages 5-15) were tested twice by the same examiner, and 10 pediatric physical therapists rated 10 randomly chosen sessions. PBS showed high test-retest (ICC = 0.998) and interrater reliability (ICC = 0.997), confirming its effectiveness as a reliable balance assessment tool
TGMD-2 (Test of Gross Motor Development-2) | baseline
  The Test of Gross Motor Development-Second Edition (TGMD-2) evaluates children's motor skills. A study assessed the Portuguese version for clarity, validity, and reliability. Two trials per child were video recorded for analysis. The motor tasks were found clear and reflective of motor development. The test showed good validity (Chi-square/df = 3.38; GFI = 0.95; AGFI = 0.92; TLI = 0.83) and strong reliability (locomotor: r = 0.82; object control: r = 0.88).
kinovea software | baseline
  Kinovea is a non-invasive, cost-effective tool for assessing thoracic kyphosis and lumbar lordosis. In a study with 18 participants, its measurements were compared to Cobb's method. Inter- and intra-rater reliability showed moderate to perfect agreement (ICC < 0.001). Validity for thoracic kyphosis was moderate and dependent on evaluator expertise, while lumbar lordosis showed weaker correlation. Kinovea proves useful for clinical and research-based postural assessments

CONTACTS AND LOCATIONS:
Overall Officials: Mahrukh Fatima, MS-PPT, Principal Investigator — Riphah International University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yuan R, Zhang J, Song P, Qin L. The relationship between screen time and gross motor movement: A cross-sectional study of pre-school aged left-behind children in China. PLoS One. 2024 Apr 5;19(4):e0296862. doi: 10.1371/journal.pone.0296862. eCollection 2024. PMID 38578800